CLINICAL TRIAL: NCT05626127
Title: Evaluation of a MRI-based Clinico-radiomics Model in Predicting Lymph Node Metastasis Status of Hilar Cholangiocarcinoma Patients: a Prospective Diagnostic Study
Brief Title: MRI-based Clinico-radiomics Predicting Lymph Node Metastasis Status of Hilar Cholangiocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-267-01
Record Dates: First submitted 2022-11-16; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: Hilar Cholangiocarcinoma; Lymph Node Metastasis; Radiomics; Machine-learning; Prognosis
MeSH Terms: conditions — Klatskin Tumor; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University: The cohort of Sun Yat-Sen Memorial Hospital of Sun Yat-sen University is the validation cohort.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — As this is a observational study, there are no interventions.

SUMMARY:
This is a prospective, observational diagnostic study aiming to assess multiparametric MRI-based clinico-radiomics for identifying lymph node metastasis status in hilar cholangiocarcinoma.

DETAILED DESCRIPTION:
A preoperative tool capable of predicting lymph node metastasis status in hilar cholangiocarcinoma is lacking and urgently needed for clinical practice. This study proposes to establish and evaluate a machine-learning algorithms of multiparametric MRI-based clinico-radiomics for identifying lymph node metastasis status in hilar cholangiocarcinoma. This study will investigate the relationship between radiomic depth information and tumor biological characteristics. The study includes the construction of capable MRI-based clinico-radiomics prediction model and the validation of the prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign an informed consent form;
2. Age 18-75 years old, both male and female;
3. ECOG performance status score (PS score) 0-2;
4. Hilar cholangiocarcinoma with resectable tumor lesions;
5. Complete the upper abdomen MRI examination before treatment;

Exclusion Criteria:

1. Accompanied with other primary malignant tumors;
2. Patients who have neoadjuvant chemotherapy or other tumor-targeted therapies;
3. Incomplete imaging or medical history data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had resectable hilar cholangiocarcinoma and completed the upper abdomen MRI examination before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastasis status | Baseline
  The value of multiparametric MRI-based clinico-radiomics in predicting lymph node metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No